CLINICAL TRIAL: NCT02353871
Title: A Phase III, Double Blind, Randomised, Placebo Controlled Study To Assess The Efficacy And Safety Of A Single Treatment Of Clostridium Botulinum Toxin Type A To Improve The Appearance Of Moderate To Severe Glabellar Lines
Brief Title: Efficacy and Safety of Clostridium Botulinum Toxin Type A to Improve Appearance of Moderate to Severe Glabellar Lines
Acronym: BTX-A-HAC NG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-52-52120-189; 2013-002321-34 (EudraCT Number)
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Moderate to Severe Glabellar Lines
Keywords: Moderate to Severe
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BTX-A-HAC NG (Experimental): Clostridium Botulinum Toxin Type A (BTX-A-HAC NG) 50 Unit (U) solution, single dose (intramuscular injection). The total treatment volume (0.25 mL) was divided into five injections (0.05 mL per injection) injected in five predefined sites across the glabellar region. A total of 50 U was injected.
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator): Single dose (intramuscular injection). The total placebo volume (0.25 mL) was divided into five injections (0.05 mL per injection) injected in five predefined sites across the glabellar region.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — A solution containing 50 U in 0.25 mL (200 U/mL). Each vial contained 0.625 mL of deliverable volume of solution. A volume of 0.25 mL, containing 50 U of BTX-A-HAC NG (i.e. 10 U/0.05 mL) was withdrawn from the vial into a syringe for administration. The total treatment volume (0.25 mL) was divided into five injections (0.05 mL per injection), each of which was to be administered into predefined sites across the glabellar region (two injections into each corrugator muscle and one injection into the procerus muscle).
  Other Names: BTX-A-HAC NG
  Arms: BTX-A-HAC NG
Drug: Placebo — A solution containing only the excipients of BTX-A-HAC NG (identical in appearance to the active product). Each vial contained 0.625 mL of deliverable volume of solution. A volume of 0.25 mL was withdrawn from the vial into a syringe for administration. The total treatment volume (0.25 mL) was divided into five injections (0.05 mL per injection), each of which was to be administered into predefined sites across the glabellar region (two injections into each corrugator muscle and one injection into the procerus muscle).
  Arms: Placebo

SUMMARY:
The purpose of this study was to demonstrate the safety and the efficacy of a single treatment of an injectable liquid form of Clostridium botulinum toxin type A haemagglutinin complex (BTX-A-HAC; hereafter referred to as BTX-A-HAC Next Generation (BTX-A-HAC NG)), used for the improvement in the appearance of moderate to severe glabellar lines (the lines between the eyebrows).

DETAILED DESCRIPTION:
At the Baseline Visit (Day 1), subjects were randomised in a ratio of 2:1 to receive either BTX-A-HAC NG solution (50 U) or placebo. Randomisation was stratified according to gender and severity of glabellar lines at maximum frown (moderate to severe) at Baseline. A single dose of BTX-A-HAC NG solution 50 U or placebo was injected on Day 1. Subjects were then monitored at the study centre for 30 minutes. On Day 4, subjects were contacted by telephone for adverse event monitoring and to record concomitant medications and treatments.

Subjects attended follow-up visits at the study centre on Days 8, 15, 29, 57, 85, 113, 148 and 183. The Day 183 follow-up visit was the end of study visit; all subjects who had completed the Day 183 Visit were considered to have completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study related procedures.
2. Male or female between 18 and 65 years of age, inclusive.
3. Had moderate or severe (Grade 2 or 3) vertical glabellar lines at maximum frown at baseline (Day 1), as assessed by the ILA using a validated 4-point photographic scale.
4. Had moderate or severe (Grade 2 or 3) vertical glabellar lines at maximum frown at baseline (Day 1), as assessed by the SSA using a validated 4-point categorical scale.
5. Were dissatisfied or very dissatisfied (Grade 2 or 3) with their glabellar lines at baseline (Day 1), as assessed by the subject's level of satisfaction.
6. Had a negative pregnancy test (for females of childbearing potential only). Nonchildbearing potential was defined as post menopausal for at least 1 year, surgical sterilisation at least 3 months before entering the study, or hysterectomy.
7. Had both the time and the ability to complete the study and comply with study instructions.

Exclusion Criteria:

1. Previous treatment with any serotype of botulinum toxin (BTX).
2. Any prior treatment with permanent fillers in the upper face including the glabellar lines area.
3. Any prior treatment with long lasting dermal fillers in the upper face including the glabellar lines area within the past 3 years and/or skin abrasions/resurfacing (whatever the interventional technic used) within the past 5 years, or photorejuvenation or skin/vascular laser intervention within the past 12 months.
4. Any planned facial cosmetic surgery during the study.
5. A history of eyelid blepharoplasty or brow lift within the past 5 years.
6. An inability to substantially reduce glabellar lines by physically spreading them apart or lack of capacity to frown.
7. An active infection or other skin problems in the upper face including the glabellar lines area (e.g. acute acne lesions or ulcers).
8. Use of concomitant therapy which, in the Investigator's opinion, would have interfered with the evaluation of the safety or efficacy of the study treatment, including medications affecting bleeding disorders (antiplatelet agents and/or anticoagulants given for treatment or prevention of cardiovascular/cerebrovascular diseases).
9. Pregnant women, nursing mothers, or women who were planning a pregnancy during the study, or believed they may be pregnant at the start of the study. Throughout the course of the study, women of childbearing potential had to use a reliable form of contraception (e.g. oral contraceptives for more than 12 consecutive weeks, or spermicide and condoms).
10. A history of drug or alcohol abuse.
11. Treatment with an experimental drug or use of any experimental device within 30 days prior to the start of the study and during the conduct of the study.
12. Known allergy or hypersensitivity to any serotype of BTX or any component of BTX-A-HAC NG.
13. Clinically diagnosed significant anxiety disorder, or any other significant psychiatric disorder (e.g. depression) that might interfere with the subject's participation in the study.
14. Use of medications that affect neuromuscular transmission, such as curare like nondepolarising agents, lincosamides, polymyxins, anticholinesterases and aminoglycoside antibiotics, within the past 30 days.
15. A history of facial nerve palsy.
16. Marked facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin.
17. The presence of any other condition (e.g. neuromuscular disorder or other disorder that could interfere with neuromuscular function), laboratory finding or circumstance that, in the judgement of the Investigator, might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (9):
- France (4):
  - Nouvelle Clinique Bel Air, Bordeaux
  - Cabinet Medical, Cannes
  - Mediti, Juan-les-Pins
  - Clinique IENA, Paris
- Germany (5):
  - Rzany & Hund Privatpraxis für Dermatologie, Berlin
  - Medical Skin Center, Düsseldorf
  - University of Hamburg, Hamburg
  - Rote Kreuz Krankenhaus, Kassel
  - Hautzentrum am Starnberger See, Starnberg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Hilton S, Kestemont P, Sattler G, Volteau M, Thompson C, Andriopoulos B, Prygova I, Berg AK, Ascher B. Liquid AbobotulinumtoxinA: Pooled Data From Two Double-Blind, Randomized, Placebo-Controlled Phase III Studies of Glabellar Line Treatment. Dermatol Surg. 2022 Nov 1;48(11):1198-1202. doi: 10.1097/DSS.0000000000003594. Epub 2022 Oct 7. PMID 36206385

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from nine active sites in France and Germany from January 2015. The study was completed in August 2015.
Pre-assignment Details: Overall, 190 subjects were screened, five of whom were screening failures. A total of 185 subjects were randomised to receive treatment. One of the subjects who was randomised to placebo did not receive study treatment due to violation of inclusion criterion 3.
Groups:
- BTX-A-HAC NG Solution (50 U): Clostridium Botulinum Toxin Type A (BTX-A-HAC NG) 50 U solution, single dose (intramuscular injection). The total treatment volume (0.25 mL) was divided into five injections (0.05 mL per injection) injected in five predefined sites across the glabellar region. A total of 50 U was injected.
- Placebo: Placebo single dose (intramuscular injection). The total placebo volume (0.25 mL) was divided into five injections (0.05 mL per injection) injected in five predefined sites across the glabellar region.
Period: Overall Study
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Started | 125 (Randomised.) | 60 (Randomised. Included a subject who was randomised by mistake (excluded from mITT population).)
Completed | 122 | 51
Not Completed | 3 | 9
Not completed — Protocol deviation | 0 | 1
Not completed — Consent withdrawn | 1 | 8
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomised population.
Groups:
- Total: Total of all reporting groups
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo | Total
Number analyzed (Participants) | 125 | 60 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (9.75) | 48.0 (9.09) | 47.8 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 52 | 160
  Male | 17 | 8 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 125 | 60 | 185
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 124 | 59 | 183
  Black/African American | 0 | 1 | 1
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Responders at Day 29 in the ILA of Glabellar Lines at Maximum Frown.
Description: ILA
  4-point photographic scale: None - Grade 0; mild - Grade 1; moderate - Grade 2; severe - Grade 3.
  A responder at maximum frown was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at maximum frown on Day 29 and a severity grade of moderate (Grade 2) or severe (Grade 3) at Baseline (Day 1).
  The adjusted proportion of responders in each treatment group was provided using a multivariate logistic regression model.
Time Frame: Day 29
Population: Modified intent-to-treat (mITT) population included all randomised subjects who received at least one injection of study treatment into one injection site and who had both Baseline and at least one postbaseline value for the ILA of glabellar lines at maximum frown. Subjects who did not have available data at Day 29 were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of responders
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Number analyzed (Participants) | 124 | 58
Adjusted percentage of responders | 88.3 [76.1 to 94.7] | 1.4 [0.3 to 6.5]
Statistical Analysis 1: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 29; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; Multivariate model, controlling for centre and stratification factors (i.e. gender and baseline ILA (maximum frown)) as fixed effects

2. Secondary Outcome: The Proportion of Responders at Each Post-treatment Visit to the Study Centre (Except Day 29) as Measured by the ILA at Maximum Frown.
Description: ILA
  4-point photographic scale: None - Grade 0; mild - Grade 1; moderate - Grade 2; severe - Grade 3.
  A responder at maximum frown was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at maximum frown at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) at Baseline (Day 1).
  The adjusted proportion of responders in each treatment group was provided using a multivariate logistic regression model.
Time Frame: Day 8, 15, 57, 85, 113, 148 and 183
Population: mITT: all randomised subjects who received at least one injection of study treatment into one injection site and who had both Baseline and at least one postbaseline value for the ILA of glabellar lines at maximum frown. N'=number of subjects with available data at the given visit; P=placebo.
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of responders
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Number analyzed (Participants) | 125 | 59
Adjusted percentage of responders
  Day 8: number analyzed (Participants) | 124 | 57
  Day 8 | 80.5 [65.3 to 90.0] | 1.3 [0.3 to 6.2]
  Day 15: number analyzed (Participants) | 124 | 59
  Day 15 | 87.0 [74.5 to 93.9] | 1.5 [0.3 to 7.0]
  Day 57: number analyzed (Participants) | 124 | 58
  Day 57 | 77.4 [63.0 to 87.3] | 1.0 [0.2 to 5.4]
  Day 85: number analyzed (Participants) | 121 | 57
  Day 85 | 51.3 [35.1 to 67.3] | 1.0 [0.2 to 5.6]
  Day 113: number analyzed (Participants) | 123 | 56
  Day 113 | 34.0 [20.5 to 50.7] | 0.8 [0.1 to 5.1]
  Day 148: number analyzed (Participants) | 121 | 51
  Day 148 | 17.1 [7.9 to 33.1] | 1.8 [0.3 to 9.8]
  Day 183: number analyzed (Participants) | 122 | 51
  Day 183 | 4.9 [0.9 to 23.2] | 0.9 [0.1 to 8.9]
Statistical Analysis 1: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA at Day 8 - BTX-A-HAC NG solution (50 U) versus placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA at Day 15 - BTX-A-HAC NG solution (50 U) versus placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA at Day 57 - BTX-A-HAC NG solution (50 U) versus placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA at Day 85 - BTX-A-HAC NG solution (50 U) versus placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA at Day 113 - BTX-A-HAC NG solution (50 U) versus placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA at Day 148 - BTX-A-HAC NG solution (50 U) versus placebo; Test type: Superiority or Other; p = 0.0035, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA at Day 183 (End of Study) - BTX-A-HAC NG solution (50 U) versus placebo; Test type: Superiority or Other; p = 0.0441, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: The Proportion of Responders on Day 29 Who Remained Responders on Days 57, 85, 113, 148 and 183 as Measured by the ILA at Maximum Frown.
Description: ILA
  4-point photographic scale: None - Grade 0; mild - Grade 1; moderate - Grade 2; severe - Grade 3.
  A responder at maximum frown was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at maximum frown at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) at Baseline (Day 1). Subjects who were not responders at Day 29 were excluded from the analysis.
  The adjusted proportion of responders in each treatment group was provided using a multivariate logistic regression model.
Time Frame: Day 57, 85, 113, 148 and 183
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of responders
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Number analyzed (Participants) | 125 | 59
Adjusted percentage of responders
  Day 57: number analyzed (Participants) | 112 | 2
  Day 57 | 87.3 [72.4 to 94.8] | 47.0 [2.8 to 96.5]
  Day 85: number analyzed (Participants) | 109 | 2
  Day 85 | 61.1 [42.5 to 77.0] | 4.9 [0.1 to 73.4]
  Day 113: number analyzed (Participants) | 111 | 2
  Day 113 | 39.6 [23.9 to 57.9] | 24.0 [0.7 to 93.5]
  Day 148: number analyzed (Participants) | 109 | 2
  Day 148 | 20.1 [9.0 to 39.0] | 32.1 [1.8 to 92.6]
  Day 183: number analyzed (Participants) | 110 | 2
  Day 183 | 5.3 [0.9 to 26.6] | 8.0 [0.2 to 76.9]
Statistical Analysis 1: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of the proportion of responders on Day 29 who remained responders at Day 57 - BTX-A-HAC NG solution (50 U) versus Placebo; Test type: Superiority or Other; p = 0.2422, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of the proportion of responders on Day 29 who remained responders at Day 85 - BTX-A-HAC NG solution (50 U) versus Placebo; Test type: Superiority or Other; p = 0.0917, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of the proportion of responders on Day 29 who remained responders at Day 113 - BTX-A-HAC NG solution (50 U) versus Placebo; Test type: Superiority or Other; p = 0.7064, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of the proportion of responders on Day 29 who remained responders at Day 148 - BTX-A-HAC NG solution (50 U) versus Placebo; Test type: Superiority or Other; p = 0.7010, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of the proportion of responders on Day 29 who remained responders at Day 183 - BTX-A-HAC NG solution (50 U) versus Placebo; Test type: Superiority or Other; p = 0.7894, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: The Proportion of Responders at Each Post-treatment Visit to the Study Centre as Measured by the ILA at Rest.
Description: ILA
  4-point photographic scale: None - Grade 0; mild - Grade 1; moderate - Grade 2; severe - Grade 3.
  A responder at rest was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at rest at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) at Baseline (Day 1).
  The adjusted proportion of responders in each treatment group was provided using a multivariate logistic regression model.
Time Frame: Day 8, 15, 29, 57, 85, 113, 148 and 183
Population: mITT: all randomised subjects who received at least one injection of study treatment into one injection site and who had both Baseline and at least one postbaseline value for the ILA of glabellar lines at maximum frown. N'=number of subjects with available data at the given visit.; P=placebo.
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of responders
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Number analyzed (Participants) | 125 | 59
Adjusted percentage of responders
  Day 8: number analyzed (Participants) | 53 | 31
  Day 8 | 73.2 [38.4 to 92.3] | 2.0 [0.2 to 15.8]
  Day 15: number analyzed (Participants) | 53 | 32
  Day 15 | 74.5 [37.7 to 93.3] | 1.3 [0.1 to 12.7]
  Day 29: number analyzed (Participants) | 53 | 32
  Day 29 | 81.1 [46.5 to 95.5] | 1.5 [0.1 to 14.4]
  Day 57: number analyzed (Participants) | 53 | 32
  Day 57 | 77.2 [41.7 to 94.1] | 0.5 [0.0 to 10.6]
  Day 85: number analyzed (Participants) | 53 | 32
  Day 85 | 58.5 [24.0 to 86.2] | 0.5 [0.0 to 8.0]
  Day 113: number analyzed (Participants) | 53 | 31
  Day 113 | 74.7 [43.5 to 91.8] | 4.8 [0.8 to 24.6]
  Day 148: number analyzed (Participants) | 51 | 29
  Day 148 | NA [NA to NA] — Not calculable due to quasi-complete separation of data point. Therefore statistical analysis was not possible. | NA [NA to NA] — Not calculable due to quasi-complete separation of data point. Therefore statistical analysis was not possible.
  Day 183: number analyzed (Participants) | 53 | 29
  Day 183 | 56.0 [26.4 to 81.9] | 10.4 [2.2 to 37.9]
Statistical Analysis 1: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 8; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; Multivariate model, controlling for centre and stratification factors (i.e. gender and baseline ILA (at rest)) as fixed effects
Statistical Analysis 2: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 15; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 29; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 57; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 85; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 113; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 183; Test type: Superiority or Other; p = 0.0015, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: The Proportion of Subjects With a Reduction of Two or More Grades in the Severity of Glabellar Lines at Each Post-treatment Visit to the Study Centre as Measured by the ILA at Maximum Frown.
Description: ILA
  4-point photographic scale: None - Grade 0; mild - Grade 1; moderate - Grade 2; severe - Grade 3.
  Adjusted proportion of subjects with a reduction of two or more grades in the severity of glabellar lines at each post-treatment visit compared with Baseline.
  The adjusted proportion of responders in each treatment group was provided using a multivariate logistic regression model.
Time Frame: Day 8, 15, 29, 57, 85, 113, 148 and 183
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of responders
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Number analyzed (Participants) | 125 | 59
Adjusted percentage of responders
  Day 8: number analyzed (Participants) | 124 | 57
  Day 8 | 56.2 [37.1 to 73.6] | 0.2 [0.0 to 3.0]
  Day 15: number analyzed (Participants) | 124 | 59
  Day 15 | 69.7 [52.0 to 83.0] | 0.2 [0.0 to 3.1]
  Day 29: number analyzed (Participants) | 124 | 58
  Day 29 | 63.6 [46.4 to 77.9] | 0.1 [0.0 to 1.8]
  Day 57: number analyzed (Participants) | 124 | 58
  Day 57 | 48.0 [31.6 to 64.9] | 0.1 [0.0 to 2.6]
  Day 85: number analyzed (Participants) | 121 | 57
  Day 85 | 24.3 [13.4 to 39.9] | 0.3 [0.0 to 4.8]
  Day 113: number analyzed (Participants) | 123 | 56
  Day 113 | 10.1 [4.3 to 21.7] | 0.3 [0.0 to 4.4]
  Day 148: number analyzed (Participants) | 121 | 51
  Day 148 | 3.5 [0.8 to 13.5] | 0.3 [0.0 to 5.4]
  Day 183: number analyzed (Participants) | 122 | 51
  Day 183 | 3.4 [0.8 to 12.6] | 1.3 [0.1 to 12.0]
Statistical Analysis 1: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 8; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 15; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 29; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 57; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 85; Test type: Superiority or Other; p = 0.0008, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 113; Test type: Superiority or Other; p = 0.0065, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 148; Test type: Superiority or Other; p = 0.0643, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of ILA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 183; Test type: Superiority or Other; p = 0.3670, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: The Proportion of Responders at Each Post-treatment Visit to the Study Centre as Measured by the Subject's Self-assessment (SSA) at Maximum Frown.
Description: SSA
  4-point photographic scale: No wrinkles - 0; Mild wrinkles - 1; Moderate wrinkles - 2; Severe wrinkles - 3.
  A responder at maximum frown was defined as having a severity grade of no wrinkles (Grade 0) or mild wrinkles (Grade 1) at maximum frown at a given visit and a severity grade of moderate wrinkles (Grade 2) or severe wrinkles (Grade 3) at Baseline (Day 1).
  The adjusted proportion of responders in each treatment group was provided using a multivariate logistic regression model.
Time Frame: Day 8, 15, 29, 57, 85, 113, 148 and 183
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of responders
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Number analyzed (Participants) | 125 | 59
Adjusted percentage of responders
  Day 8: number analyzed (Participants) | 124 | 57
  Day 8 | 62.0 [47.2 to 74.9] | 5.1 [1.6 to 14.8]
  Day 15: number analyzed (Participants) | 124 | 59
  Day 15 | 75.6 [61.8 to 85.6] | 4.4 [1.3 to 13.7]
  Day 29: number analyzed (Participants) | 124 | 58
  Day 29 | 76.0 [62.2 to 85.9] | 5.2 [1.7 to 15.0]
  Day 57: number analyzed (Participants) | 124 | 58
  Day 57 | 67.5 [52.4 to 79.6] | 2.2 [0.6 to 8.3]
  Day 85: number analyzed (Participants) | 121 | 57
  Day 85 | 61.8 [46.1 to 75.3] | 3.9 [1.1 to 12.6]
  Day 113: number analyzed (Participants) | 123 | 56
  Day 113 | 46.2 [32.8 to 60.2] | 9.8 [3.9 to 22.5]
  Day 148: number analyzed (Participants) | 121 | 51
  Day 148 | 44.1 [31.2 to 57.7] | 13.1 [5.3 to 28.9]
  Day 183: number analyzed (Participants) | 122 | 51
  Day 183 | 27.0 [16.4 to 41.1] | 6.0 [1.8 to 17.8]
Statistical Analysis 1: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of SSA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 8; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of SSA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 15; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of SSA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 29; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of SSA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 57; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of SSA - Dysport 50 U versus Placebo at Day 85; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of SSA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 113; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of SSA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 148; Test type: Superiority or Other; p = 0.0011, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of SSA - BTX-A-HAC NG solution (50 U) versus Placebo at Day 183; Test type: Superiority or Other; p = 0.0036, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: The Proportion of Responders at Each Post-treatment Visit to the Study Centre as Measured by the Subject's Level of Satisfaction With the Appearance of Their Glabellar Lines.
Description: Adjusted proportion of responders at each post-treatment visit (measured by the subject's level of satisfaction with the appearance of their glabellar lines).
  4-point categorical scale: Grade 0 - very satisfied; Grade 1 - satisfied; Grade 2 - dissatisfied; Grade 3 - very dissatisfied.
  A responder was defined as having a satisfaction rating of very satisfied (Grade 0) or satisfied (Grade 1) at a given visit and a satisfaction rating of dissatisfied (Grade 2) or very dissatisfied (Grade 3) at Baseline (Day 1).
  The adjusted proportion of responders in each treatment group was provided using a multivariate logistic regression model.
Time Frame: Day 8, 15, 29, 57, 85, 113, 148 and 183
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of responders
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Number analyzed (Participants) | 125 | 59
Adjusted percentage of responders
  Day 8: number analyzed (Participants) | 124 | 57
  Day 8 | 72.7 [58.9 to 83.2] | 4.9 [1.6 to 14.5]
  Day 15: number analyzed (Participants) | 124 | 59
  Day 15 | 80.6 [68.4 to 88.9] | 7.9 [3.1 to 19.1]
  Day 29: number analyzed (Participants) | 124 | 58
  Day 29 | 80.9 [68.7 to 89.1] | 8.3 [3.1 to 20.2]
  Day 57: number analyzed (Participants) | 124 | 58
  Day 57 | 74.7 [61.2 to 84.6] | 5.9 [2.1 to 15.3]
  Day 85: number analyzed (Participants) | 121 | 57
  Day 85 | 70.9 [56.1 to 82.3] | 7.3 [2.7 to 18.7]
  Day 113: number analyzed (Participants) | 123 | 56
  Day 113 | 61.9 [48.3 to 73.8] | 9.8 [4.0 to 22.2]
  Day 148: number analyzed (Participants) | 121 | 51
  Day 148 | 58.9 [45.4 to 71.3] | 12.3 [5.0 to 27.3]
  Day 183: number analyzed (Participants) | 122 | 51
  Day 183 | 49.8 [36.3 to 63.3] | 11.3 [4.5 to 25.6]
Statistical Analysis 1: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of subject's level of satisfaction - BTX-A-HAC NG solution (50 U) versus Placebo at Day 8; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of subject's level of satisfaction - BTX-A-HAC NG solution (50 U) versus Placebo at Day 15; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of subject's level of satisfaction - BTX-A-HAC NG solution (50 U) versus Placebo at Day 29; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of subject's level of satisfaction - BTX-A-HAC NG solution (50 U) versus Placebo at Day 57; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of subject's level of satisfaction - BTX-A-HAC NG solution (50 U) versus Placebo at Day 85; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of subject's level of satisfaction - BTX-A-HAC NG solution (50 U) versus Placebo at Day 113; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of subject's level of satisfaction - BTX-A-HAC NG solution (50 U) versus Placebo at Day 148; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of subject's level of satisfaction - BTX-A-HAC NG solution (50 U) versus Placebo at Day 183; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical tests were two-sided with a type I error rate at 5%; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: The Time to Onset of Treatment Response Based on the Subject's Diary Card.
Description: Median time to onset of treatment response: subjects asked to record their assessment of study treatment response in a diary card on Days 1 to 7. They responded 'yes' or 'no' to the following question: 'since being injected have you noticed an improvement in the appearance of your glabellar lines (lines between your eyebrows)?'
Time Frame: Day 1 to 7
Population: mITT: All randomised subjects who received at least one injection of study treatment into one injection site and who had both Baseline and at least one postbaseline value for the ILA of glabellar lines at maximum frown. One subject from the placebo group was excluded from the analysis due to missing data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Number analyzed (Participants) | 125 | 58
Days | 3.0 [2.0 to 3.0] | NA [NA to NA] — Median could not be calculated because insufficient number of participants with events in the placebo group (11 events).
Statistical Analysis 1: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of time to onset of treatment response - BTX-A-HAC NG solution (50 U) versus Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: BTX-A-HAC NG Solution (50 U) vs Placebo; Comparison of time to onset of treatment response - BTX-A-HAC NG solution (50 U) versus placebo; Test type: Superiority or Other; p < 0.0001, Cox proportional hazard model; Centre, gender and ILA baseline severity score used as covariates; Hazard Ratio (HR) = 6.561

ADVERSE EVENTS:
Time Frame: Screening until end of study (Day 183)/early withdrawal
Description: Adverse events were elicited by direct, nonleading questioning or by spontaneous reports. An adverse event was defined as the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Arm/Group | BTX-A-HAC NG Solution (50 U) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/125 | 1/59
Other Adverse Events (participants affected / at risk) | 49/125 | 17/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTX-A-HAC NG Solution (50 U) (N=125) | Placebo (N=59)
Mydriasis (Eye disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTX-A-HAC NG Solution (50 U) (N=125) | Placebo (N=59)
Nasopharyngitis (Infections and infestations) | 10 (10) | 5 (6)
Influenza (Infections and infestations) | 3 (4) | 3 (3)
Headache (Nervous system disorders) | 18 (27) | 2 (2)
Injection site pain (General disorders) | 10 (10) | 3 (3)
Tonsillitis (Infections and infestations) | 3 (3) | 0 (0)
Brow ptosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0)
Eyelid oedema (Eye disorders) | 2 (2) | 0 (0)
Blepharochalasis (Eye disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritis generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Median could not be calculated because insufficient number of participants with events in the placebo group (3 events for ILA and 8 for SSA).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A plan for scientific publication and presentation of the results could be agreed and implemented by the study investigators or a steering committee. The sponsor required that reasonable opportunity be given to review the content and conclusions of any abstract, presentation, or paper before the material was submitted for publication or communicated. This condition also applied to any amendments that were subsequently requested by referees or journal editors.